CLINICAL TRIAL: NCT02783443
Title: Effect General and Regional Anesthesia on Glycocalyx
Status: Completed | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Vladimir Cerny, prof. Vladimir Cerny, MD, PhD, FCCM, University Hospital Hradec Kralove
Other Study IDs: AZVCR 9307_2
Record Dates: First submitted 2016-05-20; First posted 2016-05-26 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Anesthesia; Glycocalyx; Perfused Boundary Region
Keywords: Anesthesia, glycocalyx, perfused boundary region
MeSH Terms: interventions — Anesthesia, General; Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- General anesthesia: Adult patients ASA 2-3 undergoing elective total knee replacement surgery under general anaesthesia.
  Interventions: Other: General anesthesia
- Regional anesthesia: Adult patients ASA 2-3 undergoing elective total knee replacement surgery under regional anaesthesia.
  Interventions: Other: Regional anesthesia

INTERVENTIONS:
Other: General anesthesia — General anesthesia
  Groups: General anesthesia
Other: Regional anesthesia — Regional anesthesia
  Groups: Regional anesthesia

SUMMARY:
Observational study evaluating effect general or regional anaesthesia on glycocalyx by using perfused Boundary Region in sublingual microcirculation.

DETAILED DESCRIPTION:
Study II: Effect general and regional anaesthesia on GCX Hypothesis to be tested: Regional anaesthesia affects GCX less than general anaesthesia.

The aim of the study: Comparison of two anaesthesia techniques with respect to GCX.

Type of the study: Observational. Subjects: Adult patients ASA 2-3 undergoing elective total knee replacement surgery under general or regional anaesthesia. Sample size calculation (based on expected difference in PRB, alpha error I = 0,05 and study power = 0,99) = 52 patients. Investigators plan to enroll of 60 consecutive patients to reach 30 patients with each type of anaesthesia. Intervention: none. Data to be recorded and analysed: Demographics, ASA, physiologic functions (during surgery and 24 hours after surgery), fluids given, sublingual microcirculation by SDF imaging will be recorded at time points: before anaesthesia, 24 hours after anaesthesia, clinical outcome indicators, microcirculatory data and Perfused Boundary Region.

ELIGIBILITY:
Inclusion Criteria:

Adult patients ASA 2-3 undergoing elective total knee replacement surgery

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients ASA 2-3 undergoing elective total knee replacement surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-06; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Cerny, MD, Principal Investigator — University Hospital Hradec Kralova, Czech Republic

IPD SHARING:
Plan to Share IPD: Yes
On request if privacy guaranteed

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | General Anesthesia | Regional Anesthesia
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Anesthesia | Regional Anesthesia | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (7) | 67 (9) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 14 | 16 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 30 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Czechia | 30 | 30 | 60
Baseline PBR [Mean (Standard Deviation); unit: micrometer] — PBR is perfused boundary region of the sublingual microcirculation as an indirect assessment of the endothelial glycocalyx thickness.
  micrometer | 2.02 (0.26) | 1.95 (0.24) | 1.99 (0.25)

OUTCOME MEASURES:

1. Primary Outcome: Change in Perfused Boundary Region (PBR)
Description: PBR is an indirect measure of glycocalyx thickness
Time Frame: Change from baseline PBR at 24 hours after surgery
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | General Anesthesia | Regional Anesthesia
Number analyzed (Participants) | 30 | 30
micrometer | 2.20 (0.25) | 2.09 (0.19)

ADVERSE EVENTS:
Time Frame: 1 year
Description: A serious adverse event represents a situation that required patient transport to the ICU or prolongation of stay in the hospital. The other adverse event represents a situation in which a doctor had been called but with no impact on patient stay or short-term outcome.
Arm/Group | General Anesthesia | Regional Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 12/30 | 1/30
Other Adverse Events (participants affected / at risk) | 12/30 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | General Anesthesia (N=30) | Regional Anesthesia (N=30)
PONV (Gastrointestinal disorders) | 8 (8) | 0 (0)
anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
obstipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
delirium (Nervous system disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | General Anesthesia (N=30) | Regional Anesthesia (N=30)
pain (Nervous system disorders) | 12 (12) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT02783443/Prot_SAP_000.pdf